CLINICAL TRIAL: NCT01123330
Title: Detroit Research Center on Oral Health Disparities
Brief Title: Evaluation of a Brief Tailored Motivational Intervention to Prevent Early Childhood Caries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Amid I. Ismail, Temple University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U54DE1426101
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Motivational Interviewing plus DVD (Experimental): Caregivers watched a 15-minute educational video designed for the project emphasizing the importance of good oral health in children, and how the caregiver can keep children free from tooth decay. The MI interviewer engaged the parent in a discussion of their thoughts and concerns regarding their child's oral health and what changes they wished to make regarding monitoring their child's oral health. Feedback from the child's dental exam was also reviewed. MI+DVD caregivers received a brochure displaying a photo of their child and for those who chose to set specific goals for their child's oral health, those goals were listed on the brochure. Caregivers choosing not to set specific goals were offered a list of 10 project recommendations regarding dietary intake, oral hygiene, and dental check-ups. The session ended with a dialogue regarding possible barriers to implementing the personal plan and how the caregiver planned to overcome those barriers.
  Interventions: Behavioral: Motivational Interviewing
- DVD only (Active Comparator): Caregivers watched the same educational video. At the end of the video, caregivers were given a glossy-printed brochure displaying the project developed recommendations as well as the child's photograph. The brochure was not re-mailed, as it was for the MI+DVD group and caregivers in this condition did not receive any feedback from the dental examination regarding their child's oral health status.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing

SUMMARY:
The Detroit Dental Health Project (DDHP)aims to promote oral health and reduce disparities within the community of low-income African-American children (0-5 years) and their main caregivers (14+ years), living in the City of Detroit. The driving theme of the Project is to identify determinants and design interventions to answer the following question: why do some low-income African-American children and their main caregivers have better oral health than others who live in the same community? The Project has 3 support cores, 4 research core projects and 1 pilot study. The Project has selected a multistage random sample of African-American families living in the poorest 39 Census Tracts in the City of Detroit. A total of 1,022 families were recruited and interviewed at a community center in Detroit during the year 2 (2002). We have collected data about the social characteristics of parents, families, and neighborhoods that are associated with disparities in oral health; lead levels in saliva and blood of the caregivers; and dietary intake. All these families will be recalled in the year 4 (2004) and year 6 (2006) for longitudinal data collection. We are currently developing a tailored multi-media educational intervention (Project #3), based on data collected in the first phase (2002). The educational intervention will be administered using a randomized controlled design in year 4 (2004). Additionally, the Project is evaluating the impact on access to dental care of a state-funded experiment on utilization where Medicaid children are managed like privately insured patients (Project #4).

DETAILED DESCRIPTION:
The principal theme of the DDHP is to investigate why some African-American children and their main caregivers have better oral health than others who live in the same community. This question dictates the design of individual projects to understand the determinants of oral health disparities.

The DDHP has the following specific aims:

1. To promote oral health and reduce the disparities in oral health within the community of low-income African-American children (0-5 years) and their main caregivers living in the City of Detroit. This goal will be addressed through understanding of the social, familial, biological, and neighborhood determinants of dental caries and periodontal disease, and designing and implementing tailored interventions to target oral health knowledge and behaviors and access to dental care.
2. To develop a multidisciplinary cadre of health providers knowledgeable about oral health care and research in the City of Detroit.
3. To assist in the provision of dental care services to low-income and dentally underserved residents of the City of Detroit.

The DDHP includes three integrated research projects that are centered on one targeted population and one research project that will evaluate the impact of a state-sponsored pragmatic experiment on access to dental care and utilization of dental services (Project 4). The DDHP also includes one pilot project that aims to develop a new index for evaluating the impact of dental aesthetics on employability and social acceptance.

The research program focuses on the determinants of oral health status (dental caries and periodontal disease) of families that include at least one child less than 6 years of age at baseline (2002-2003) and the main caregiver of the child. The main caregiver is the individual who is responsible for feeding, bathing, and nurturing a child emotionally, mentally, and physically at the primary home of residence. The cohort will be followed for 4 years with a second assessment (interviews and dental examinations) in the fourth year and in the six year of the funding cycle of the DDHP.

The DDHP includes the following 4 research projects:

Project 1: Socio-cultural determinants, context of parenting and children's oral health: This project is led by Kristine Siefert, MSW, PhD, MPH, Professor, School of Social Work, University of Michigan. Dr. Siefert contends that current research is inadequate to explain the process by which social location translates into poor oral health starting in earliest childhood. Without an understanding of the process by which this occurs, preventive interventions are unlikely to succeed. Accordingly, the aim of her research is to examine the influence of material and social context at the individual (e.g., poverty and material hardship, institutional and personally mediated discrimination, and social and cultural supports and resources) and neighborhood (Census track, police precinct, and City of Detroit data) levels, on child oral health, and the mediating and moderating effects of caregiver parenting behaviors and beliefs. Using an ecosocial framework, this project focuses on identifying potent and modifiable determinants of health promotion as a part of parenting. To understand how context influences parenting and parenting influences outcomes over time, the project uses a longitudinal design, and takes advantage of newly developed techniques in growth curve and hierarchical modeling. Data from this project will provide information on interactions among social and cultural factors and caretaking behaviors of the caregivers and oral health behaviors of children and their risk of developing severe dental caries.

Project 2: Lead exposure and dietary factors in children's oral health: This project is led by Brian A. Burt, BDS, PhD, Professor, School of Public Health, University of Michigan. This study seeks to identify the relationships between lead levels, intake of dietary fats and sugars, and dental caries experienced in disadvantaged African-American children, and to identify how these variables in the caregiver relate to the child's oral health status. The purpose of this research is to identify areas for successful intervention toward reducing the disparities between those with the poorest oral health and their better-off peers. The data will be collected using a food frequency questionnaire (FFQ) and a dental examination for the caregiver and the index child. In addition, the caregiver will be asked for a finger stick blood sample and a saliva sample (for lead and other metal assay). Blood and/or saliva samples from the children will only be sought in years 4 and 6. Participants will also be measured for height and weight at the first and subsequent examinations. For testing the hypotheses, the outcomes are severe dental caries experienced in the child, and exposures are lead levels in child, and sugars and fats in the diets of child and caregiver. Other variables, such as the demographic information collected in other studies and body mass index of the caregiver and child, will be included in the multivariate analyses to determine relative risk. Nested case-control studies, with several measures of caries as the outcomes, will also be conducted. The significance of this study is that it will identify areas for intervention and produce a unique database from an African-American population. The 0-2 child's FFQ, developed for this study, will also be a valuable tool for other studies of child obesity, nutrition, and diabetes in young African Americans.

Project 3: Efficacy of a tailored oral health education program: This project will be led by David Williams PhD, Institute for Social Research and Jorge Delva PhD, School of Social Work, University of Michigan. The long-term objective of this project is to develop an effective tailored behavior change education program to promote and maintain good oral health and prevent oral diseases among low-income children and their caregivers. To achieve this, a multi-method and multi-level intervention that targets not only parental behaviors and beliefs but also contextual determinants of oral health behaviors to be identified by Project 1 will be designed. Due to the current lack of tailored self-help behavior change dental interventions, substantial time and resources are needed to develop the content and to test the instruments and feasibility of the proposed intervention. This project has five specific aims: (1) To design and produce two interventions to promote oral health and prevent oral disease among caregivers and their children: (i) an interactive, tailored, theory-driven, behavior change education program, and (ii) an untailored health information (HI) comparison program. (2) To assess the feasibility and usability of these unique interventions with a small-scale feasibility study prior their final implementation. (3) To revise the interventions based on the findings of the feasibility study and implement the efficacy trial. (4) To evaluate the efficacy of the interventions with two clinical outcomes: gingivitis among caregivers and untreated tooth decay among caregivers and their children. (5) To examine the extent to which the clinical outcomes are mediated by the affective, evaluative, and situational individual factors influenced by the tailored intervention, or by broader psychosocial factors addressed in other projects. The efficacy of the tailored intervention, whether it results in better oral health than the untailored HI intervention, will be tested in a randomized controlled trial. In year 4 of the longitudinal research, the participating caregivers will be randomly assigned to one of the two education programs at the beginning of the intervention session. The oral examination at year 4 will be the baseline measurement of this trial, and changes in the outcomes will be assessed in the follow-up examination in year 6. The research team will be masked from the assignment to the intervention regimens. Production and evaluation of a state-of-the-science, tailored multi-method, multi-level program for oral health will provide an opportunity to obtain currently non-existent information about the ability to influence behaviors that determine oral health status among low-income African American caregivers and their children.

Project 4: A pragmatic study of a new payment system for Medicaid: This study, led by Stephen A. Eklund, DDS, DrPH, School of Public Health, University of Michigan, monitors utilization of dental care in Michigan children, in order to evaluate the effectiveness of recent and future SCHIP (State Children's Health Insurance Program) and Medicaid initiatives in reducing disparities in access to and utilization of dental care. Evidence from many sources demonstrates a wide disparity in utilization of dental care that is associated with the socioeconomic status of children. Disparities exist as measured by both visits for dental care as well as untreated oral disease. Dental insurance claims data will be used to demonstrate historical patterns of utilization and the disparities between privately-insured and Medicaid-eligible children. This project specifically investigates an on-going program, funded by the State of Michigan, in which about 100,000 Medicaid children are eligible for a privately operated dental insurance program (by Delta Dental Plan of Michigan). Each Medicaid-eligible child living in 37 counties in Michigan receives a dental insurance card (the same card held by Delta Dental Plan privately insured beneficiaries) and dentists receive between 70 and 80% reimbursement for the cost of dental care. Future data from both the privately-insured child population in Michigan and from the newly-implemented private-insurance based SCHIP and Medicaid programs in Michigan will then be monitored for the next several years to assess the ability of these innovative methods of payment and administration to reduce the historical disparities in dental care utilization. Specific null hypotheses to be tested are: 1) Payment for dental care at market rates will result in no difference in the percent of children with at least one dental visit per year, among children with Medicaid, SCHIP, or private insurance coverage, 2) Payment for dental care at market rates will result in no difference in the distance traveled to receive care, among children with Medicaid, SCHIP, or private insurance coverage, and 3) Payment for dental care at market rates will result in no difference in the mix of services received among children with Medicaid, SCHIP, or private insurance coverage.

Dr. Eklund's project is the only project of the Center that is not focused on African Americans living in the 39 Census Tracts with the lowest average family income in the city. However, his research project tests an important intervention that has not yet been implemented in the Detroit area. The analysis of the Michigan experiment will provide evidence on whether policy initiatives can have an impact on access to dental care in low-income families and whether this information can be used to develop programs specific to Detroit.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* 0-5 years of age
* below 250% of poverty

Exclusion Criteria:

* None

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2042 (Actual)
Dates: Start 2001-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Carious lesions | Measures at baseline (2002-03); wave 2 (2004-05); wave 3 (2007)
  The carious process was measured using the International Caries Detection and Assessment System (ICDAS). The codes range from measurement of the first visible carious change in enamel (Code 1) to extensive cavitation (Code 6). Both primary carious lesions and lesions adjacent to restorations and sealants (CARS) were recorded,.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Delva J, Tellez M, Finlayson TL, Gretebeck KA, Siefert K, Williams DR, Ismail AI. Cigarette smoking among low-income African Americans: a serious public health problem. Am J Prev Med. 2005 Oct;29(3):218-20. doi: 10.1016/j.amepre.2005.05.004. PMID 16168872
- [Result] Delva J, Tellez M, Finlayson TL, Gretebeck KA, Siefert K, Williams DR, Ismail AI. Correlates of cigarette smoking among low-income African American women. Ethn Dis. 2006 Spring;16(2):527-33. PMID 17682259
- [Result] Finlayson TL, Siefert K, Ismail AI, Delva J, Sohn W. Reliability and validity of brief measures of oral health-related knowledge, fatalism, and self-efficacy in mothers of African American children. Pediatr Dent. 2005 Sep-Oct;27(5):422-8. PMID 16435644
- [Result] Finlayson TL, Siefert K, Ismail AI, Sohn W. Psychosocial factors and early childhood caries among low-income African-American children in Detroit. Community Dent Oral Epidemiol. 2007 Dec;35(6):439-48. doi: 10.1111/j.1600-0528.2006.00352.x. PMID 18039285
- [Result] Finlayson TL, Siefert K, Ismail AI, Sohn W. Maternal self-efficacy and 1-5-year-old children's brushing habits. Community Dent Oral Epidemiol. 2007 Aug;35(4):272-81. doi: 10.1111/j.1600-0528.2007.00313.x. PMID 17615014
- [Result] Reisine S, Ajrouch KJ, Sohn W, Lim S, Ismail A. Characteristics of African-American male caregivers in a study of oral health in Detroit--a brief communication. J Public Health Dent. 2009 Summer;69(3):197-200. doi: 10.1111/j.1752-7325.2008.00115.x. PMID 19192101
- [Result] Sanders AE, Lim S, Sohn W. Resilience to urban poverty: theoretical and empirical considerations for population health. Am J Public Health. 2008 Jun;98(6):1101-6. doi: 10.2105/AJPH.2007.119495. Epub 2008 Apr 29. PMID 18445798
- [Result] Siefert K, Finlayson TL, Williams DR, Delva J, Ismail AI. Modifiable risk and protective factors for depressive symptoms in low-income African American mothers. Am J Orthopsychiatry. 2007 Jan;77(1):113-23. doi: 10.1037/0002-9432.77.1.113. PMID 17352592
- [Result] Burt BA, Kolker JL, Sandretto AM, Yuan Y, Sohn W, Ismail AI. Dietary patterns related to caries in a low-income adult population. Caries Res. 2006;40(6):473-80. doi: 10.1159/000095645. PMID 17063017
- [Result] Kolker JL, Yuan Y, Burt BA, Sandretto AM, Sohn W, Lang SW, Ismail AI. Dental caries and dietary patterns in low-income African American children. Pediatr Dent. 2007 Nov-Dec;29(6):457-64. PMID 18254414
- [Result] Lim S, Sohn W, Burt BA, Sandretto AM, Kolker JL, Marshall TA, Ismail AI. Cariogenicity of soft drinks, milk and fruit juice in low-income african-american children: a longitudinal study. J Am Dent Assoc. 2008 Jul;139(7):959-67; quiz 995. doi: 10.14219/jada.archive.2008.0283. PMID 18594082
- [Result] Lim S, Zoellner JM, Lee JM, Burt BA, Sandretto AM, Sohn W, Ismail AI, Lepkowski JM. Obesity and sugar-sweetened beverages in African-American preschool children: a longitudinal study. Obesity (Silver Spring). 2009 Jun;17(6):1262-8. doi: 10.1038/oby.2008.656. Epub 2009 Feb 5. PMID 19197261
- [Result] Nriagu J, Burt B, Linder A, Ismail A, Sohn W. Lead levels in blood and saliva in a low-income population of Detroit, Michigan. Int J Hyg Environ Health. 2006 Mar;209(2):109-21. doi: 10.1016/j.ijheh.2005.11.005. Epub 2006 Jan 27. PMID 16443391
- [Result] Ismail AI, Sohn W, Lim S, Willem JM. Predictors of dental caries progression in primary teeth. J Dent Res. 2009 Mar;88(3):270-5. doi: 10.1177/0022034508331011. PMID 19329463
- [Result] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Result] Ismail AI, Sohn W, Tellez M, Willem JM, Betz J, Lepkowski J. Risk indicators for dental caries using the International Caries Detection and Assessment System (ICDAS). Community Dent Oral Epidemiol. 2008 Feb;36(1):55-68. doi: 10.1111/j.1600-0528.2006.00369.x. PMID 18205641
- [Result] Ismail AI, Lim S, Sohn W, Willem JM. Determinants of early childhood caries in low-income African American young children. Pediatr Dent. 2008 Jul-Aug;30(4):289-96. PMID 18767507
- [Result] Li Y, Ismail AI, Ge Y, Tellez M, Sohn W. Similarity of bacterial populations in saliva from African-American mother-child dyads. J Clin Microbiol. 2007 Sep;45(9):3082-5. doi: 10.1128/JCM.00771-07. Epub 2007 Jul 18. PMID 17634300
- [Result] Reisine S, Tellez M, Willem J, Sohn W, Ismail A. Relationship between caregiver's and child's caries prevalence among disadvantaged African Americans. Community Dent Oral Epidemiol. 2008 Jun;36(3):191-200. doi: 10.1111/j.1600-0528.2007.00392.x. PMID 18474051
- [Result] Sohn W, Ismail A, Amaya A, Lepkowski J. Determinants of dental care visits among low-income African-American children. J Am Dent Assoc. 2007 Mar;138(3):309-18; quiz 395-396, 398. doi: 10.14219/jada.archive.2007.0163. PMID 17332036
- [Result] Sohn W, Taichman LS, Ismail AI, Reisine S. Caregiver's perception of child's oral health status among low-income African Americans. Pediatr Dent. 2008 Nov-Dec;30(6):480-7. PMID 19186773
- [Result] Tellez M, Sohn W, Burt BA, Ismail AI. Assessment of the relationship between neighborhood characteristics and dental caries severity among low-income African-Americans: a multilevel approach. J Public Health Dent. 2006 Winter;66(1):30-6. doi: 10.1111/j.1752-7325.2006.tb02548.x. PMID 16570748
- [Result] Ajrouch KJ, Reisine S, Lim S, Sohn W, Ismail A. Situational stressors among African-American women living in low-income urban areas: the role of social support. Women Health. 2010 Mar;50(2):159-75. doi: 10.1080/03630241003705045. PMID 20437303
- [Result] Taichman LS, Sohn W, Lim S, Eklund S, Ismail A. Assessing patterns of restorative and preventive care among children enrolled in Medicaid, by type of dental care provider. J Am Dent Assoc. 2009 Jul;140(7):886-94. doi: 10.14219/jada.archive.2009.0282. PMID 19571052
- [Result] Ismail AI, Ondersma S, Jedele JM, Little RJ, Lepkowski JM. Evaluation of a brief tailored motivational intervention to prevent early childhood caries. Community Dent Oral Epidemiol. 2011 Oct;39(5):433-48. doi: 10.1111/j.1600-0528.2011.00613.x. Epub 2011 Mar 29. PMID 21916925